CLINICAL TRIAL: NCT07324096
Title: MC250406 Feasibility Study: Automated Risk Stratification, Serial AI-Augmented Imaging, and Biobanking for Early Detection of Sporadic Pancreatic Cancer (AI-PACED)
Brief Title: A Screening Program to Improve the Early Detection of Sporadic Pancreatic Cancer in Individuals With a High-Risk of Developing Pancreatic Cancer
Acronym: AI-PACED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MC250406; NCI-2025-09279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-009433 (Other: Mayo Clinic Institutional Review Board); MC250406 (Other: Mayo Clinic)
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; Contrast Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All CT scans obtained under the study will be interpreted by qualified radiologists who are not part of the study team and are blinded to study objectives.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A1 (CT, blood, EMR surveillance) (Experimental): Patients undergo contrast-enhanced abdominal CT and blood sample collection at baseline, 6 months, and 12 months in the absence of unacceptable toxicity. Patients also undergo EMR surveillance for PDA diagnosis for up to 36 months.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography with Contrast; Other: Electronic Health Record Review
- Group A2 (blood, EMR surveillance) (Experimental): Patients undergo blood sample collection at baseline, 6 months, and 12 months in the absence of unacceptable toxicity. Patients also undergo EMR surveillance for PDA diagnosis for up to 36 months.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review
- Group B (EMR surveillance) (Active Comparator): Patients undergo EMR surveillance for PDA diagnosis for up to 36 months.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Group A1 (CT, blood, EMR surveillance); Group A2 (blood, EMR surveillance)
Procedure: Computed Tomography with Contrast — Undergo contrast-enhanced abdominal CT
  Other Names: Contrast Enhanced Computed Tomography; CONTRAST ENHANCED CT SCAN; Contrast-enhanced Computed Tomography; CT Scan With Contrast; CT with Contrast
  Arms: Group A1 (CT, blood, EMR surveillance)
Other: Electronic Health Record Review — Undergo electronic medical record (EMR) surveillance

SUMMARY:
This clinical trial studies a new screening program to improve the early detection of sporadic pancreatic cancer in individuals with a high risk of developing pancreatic cancer. Pancreatic cancer remains one of the deadliest solid tumors, characterized by a long phase without symptoms followed by rapid progression once clinically evident. Despite advancements in treatment, the survival rate for pancreatic cancer remains low. Research has helped to identify a subset of individuals with a markedly high short-term risk for developing pancreatic cancer, which includes adults aged 50 and older with glycemically-defined new-onset diabetes and an Enriching New-Onset Diabetes for Pancreatic Cancer (ENDPAC) score ≥ 3. However, current practice guidelines do not provide clear pathways for surveillance or early detection. The screening program in this trial combines repeated contrast-enhanced computed tomography (CT) scans using artificial intelligence (AI) and blood draws. Contrast-enhanced CT is an imaging technique which creates a series of detailed pictures of areas inside the body; the pictures are created by a computer linked to an x-ray machine and a contrast agent is used to enhance the images. The images are then reviewed using AI, which may make it easier to spot cancer earlier on the CT scans than with the human eye. Studying samples of blood in the laboratory from high-risk individuals may help doctors understand more about why they may develop pancreatic cancer. This may be an effective way to screen high-risk individuals and improve the early detection of sporadic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 and ≤ 85 years
* Glycemically-defined new-onset diabetes (gNOD) with onset ≤ 180 days preceding enrollment
* Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) score ≥ 3, based on validated risk stratification models
* Provide written or remote informed consent

Exclusion Criteria:

* Prior diagnosis of pancreatic ductal adenocarcinoma (PDA)
* Known hereditary cancer syndromes (e.g., BRCA1/2, Lynch syndrome, Peutz-Jeghers)
* Prior history of pancreatic surgery
* Pancreatic cyst surveillance at time of registration
* Contraindications to contrast-enhanced CT imaging per standard clinical practice at time of registration

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment yield (Feasibility) | Up to 3 years
  Will assess the feasibility of protocol implementation as defined by recruitment yield (% of flagged high-risk individuals who consent). Descriptive statistics will be used to summarize feasibility endpoints.
Imaging adherence rates (Feasibility) | Up to 3 years
  Will assess the feasibility of protocol implementation as defined by imaging adherence rates (% completing 3 scheduled computed tomography scans). Descriptive statistics will be used to summarize feasibility endpoints.
Blood collection success rates (Feasibility) | Up to 3 years
  Will assess the feasibility of protocol implementation as defined by blood collection success rates (% completing 3 scheduled blood collections). Descriptive statistics will be used to summarize feasibility endpoints.
Completeness of electronic medical record (EMR)-based follow-up (Feasibility) | Up to 3 years
  Will assess the feasibility of protocol implementation as defined by completeness of EMR-based follow-up (% of participants with outcome ascertainment). Descriptive statistics will be used to summarize feasibility endpoints.

SECONDARY OUTCOMES:
Time from glycemically-defined new-onset diabetes (gNOD) onset to pancreatic ductal adenocarcinoma (PDA) diagnosis | Up to 3 years
  Time to PDA diagnosis will be compared between cohorts.
Proportion of PDAs diagnosed at stage 0/I | Up to 3 years
  Comparisons between cohorts will employ log-rank tests. Will also employ Cox proportional hazards models adjusted for baseline covariates (exploratory only).
Rate and type of incidental findings requiring downstream evaluation | Up to 3 years
  Comparisons between cohorts will employ log-rank tests. Will also employ Cox proportional hazards models adjusted for baseline covariates (exploratory only).
Artificial intelligence (AI)-detected imaging signatures and standard radiologist interpretations | Up to 3 years
  Will complete discordance analysis between AI-detected imaging signatures and standard radiologist interpretations, including rates of earlier detection and false positives.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit H. Goenka, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials